CLINICAL TRIAL: NCT02772029
Title: A Pilot Study of Apatinib for Advanced Hepatocellular Carcinoma Patients After First-line Treatment Failure
Brief Title: A Study of Apatinib for Advanced Hepatocellular Carcinoma Patients After First-line Treatment Failure
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Sheng Guan, Director of department of interventional neurology, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 41580193-4
Record Dates: First submitted 2016-05-10; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apatinib Mesylate Tablets (Experimental): Apatinib (Apatinib Mesylate Tablets) 750 mg is administered orally daily, until disease progression or intolerable toxicity.
  Interventions: Drug: Apatinib Mesylate Tablets

INTERVENTIONS:
Drug: Apatinib Mesylate Tablets — Apatinib 750 mg is administered orally daily, until disease progression or untolerable toxicity.
  Other Names: Apatinib

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the lethal human cancers worldwide and its incidence matches mortality, reflecting the poor prognosis of this disease. The surgical resection rate of HCC is low, and the prognosis is poor. Although transarterial chemoembolization (TACE) is the main treatment for HCC patients who are not candidates for surgical resection, it is not considered a curative procedure. For HCC, poor TACE efficacy or TACE failure may be related to tumor angiogenesis of the residual disease. Among the many regulatory factors in tumor angiogenesis, hypoxia-inducible factor-1α (HIF-1α) and vascular endothelial growth factor (VEGF) play vital roles in this process.

Sorafenib is the first systemic treatment drug, which has been approved by the FDA for advanced HCC. In order to find an new VEGFR-inhibitor with better effect and lower toxicity, Jiangsu Hengrui Medicine Co., Ltd. developed Apatinib, a high-performance VEGFR-2 tyrosine kinase inhibitor. Apatinib plays anti angiogenic effect in the treatment of malignant tumor mainly through inhibition of VEGFR-2, in vivo and in vitro experiments showed good tumor growth inhibitory activity on glioma, this study aims to further verify the efficacy and safety of Apatinib for first-line treatment failure hepatocellular carcinoma patients, the primary endpoint is time to progression(TTP).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic or cytologic diagnosis of hepatocellular carcinoma, imaging diagnosis should be compatible with chinese standard for diagnosis and treatment of primary liver cancer (Edition 2011)
* Have progressed after systematic chemotherapy/target therapy, or cannot tolerated with first-line treatment, and have at least one measurable lesion. according to RECIST 1.1, the long diameter of measurable lesion should be more or equal than 10mm, or the short diameter of a enlarged lymph node should be more or equal than 15mm, the maximum diameter of a viable tumor should be no more than 15cm
* The previous chemotherapy and the present trial registration must be at least 2 weeks apart. And they must have recovered from any toxicity of a previous chemotherapy
* Patients with Child Pugh Class A & B disease are eligible for the study
* Patients with Barcelona Clinic Liver Cancer stage B or C are eligible for the study
* Eastern Cooperative Oncology Group performance score (PS): 0-2
* Life expectancy of at least 12 weeks
* Hepatitis B virus DNA<2000 IU/ml
* Adequate organ function meeting the following:

  * Bone marrow: absolute neutrophil count ≥1.5×109/L (1500/mm3); platelet ≥ 75×109/L; hemoglobin ≥9 g/dL
  * Liver: Serum bilirubin ≤ 1.5 ×ULN, AST and ALT ≤ 5 ×ULN, ALB ≥ 29 g/L
  * Kidney: Cr ≤1.5 ×upper limit of normal
* Within 7 days prior to the start of therapy, women of child-bearing potential must undergo a pregnancy test, which must be negative; men of child-bearing potential: contraceptive measures must be adopted during treatment and within 8 weeks afterward
* Subjects who understand and voluntarily signed a written informed consent form

Exclusion Criteria:

* Diagnosed with cholangiocellular carcinoma, mixed cell carcinoma and fibrolamellar hepatocellular carcinoma
* History of other malignancy within 5 years except for non-melanoma skin cancer, cervix in situ carcinoma
* Prepared for liver transplantation
* Patients with contraindications (active bleeding, ulcers, intestinal perforation, intestinal obstruction, within 30 days after major surgery, uncontrolled high blood pressure medication, III-IV level cardiac insufficiency, severe liver and kidney dysfunction)
* A previous history of Interstitial pulmonary disease, drug-induced interstitial disease, radiation pneumonitis requiring hormonal therapy or active interstitial lung disease with any clinical evidence
* Use of CYP3A4 inhibitor within 7 days or CYP3A4 inducer within 12 days prior to enrollment
* Patients with central nervous system metastases or brain metastasis
* Previous definite diagnosis of neuropsychiatric disturbances, including epilepsy or dementia
* Pregnant or lactating women
* Patients with bone metastasis received palliative radiation within 4 weeks prior to enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
time to progression | 1 year

SECONDARY OUTCOMES:
overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: sheng guan, Principal Investigator — The First Affiliated Hospital of Zhengzhou University

IPD SHARING:
Plan to Share IPD: No